CLINICAL TRIAL: NCT02008799
Title: Intra Testicular Artery Injection of Bone Marrow Stem Cell in Management of Azoospermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Man Clinic for Andrology, Male Infertility and Sexual Dysfunction (Other)
Responsible Party: Principal Investigator, Khaled Abdulmoneim Gadalla, Prof Dr, Man Clinic for Andrology, Male Infertility and Sexual Dysfunction
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SCA2013
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Azoospermia
Keywords: Stem cell, infertility, Azoospermia
MeSH Terms: conditions — Azoospermia; Infertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone marrow stem cell injection (Experimental): through special butterfly inject stem cell in testicular artery and inside tubules
  Interventions: Procedure: Bone marrow stem cell injection

INTERVENTIONS:
Procedure: Bone marrow stem cell injection — Injection should be in testis and testicular artery

SUMMARY:
Azoospermia due to low sperm production (non-obstructive azoospermia) affects approximately 1% of the male population and 10% of men who seek fertility evaluation. Testis biopsy reveals that these men have Sertoli cell-only pattern, maturation arrest, or hypospermatogenesis. Until recently, it was assumed that men with non-obstructive azoospermia were untreatable. Indeed, these patients were often referred to as being "sterile" or having "testicular failure." We start to use stem cell in treatment of such patients by injecting the stem cell at the testis and the testicular artery in one group and at the testis only in other group

ELIGIBILITY:
Inclusion Criteria:

- Azoospermia

Exclusion Criteria:

- Absent or surgical removed testes

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Semen Analysis | Three to six months
  After stem cell injection by three to six months we evaluate the outcome by semen analysis

SECONDARY OUTCOMES:
Inhibin B Hormone | Three to six months
  If semen analysis still azoo we do Inhibin B Hormone

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Gadalla, MD, Principal Investigator — Man Clinic
Locations (1):
- Man Clinic, Cairo, Egypt